CLINICAL TRIAL: NCT07079046
Title: Efficacy of Satisens® in Reducing Emotional Eating
Acronym: Satisens
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: José Enrique de la Rubia Ortí, Ph (Other)
Collaborators: VINABAS FORMULATIONS SL (Industry)
Responsible Party: Sponsor-Investigator, José Enrique de la Rubia Ortí, Ph, Principal Investigator, Fundación Universidad Católica de Valencia San Vicente Mártir
Organization: Fundación Universidad Católica de Valencia San Vicente Mártir (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UCV/2024-2025/015
Record Dates: First submitted 2025-06-18; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Emotional Eating; Overweight or Obesity; Hormonal Changes; Neurotransmitter Agents; Food Cravings; Appetite Regulation; Body Weight; Inflammation Biomarkers
Keywords: Emotional Eating; Appetite Regulation; Food Craving; Sweet Cravings; Obesity Prevention; Dietary Supplement; Plant Extracts; Lemon Verbena; Hibiscus sabdariffa; Polyphenols; Inflammation; Nutritional Intervention; Clinical Trial; Biomarkers
MeSH Terms: conditions — Emotional Eating; Overweight; Obesity; Body Weight; Inflammation | interventions — Sucrose

STUDY DESIGN:
Intervention Model Description: This is a prospective, longitudinal, mixed-method, analytical, and experimental clinical trial. Participants will be randomly assigned to one of three groups: an intervention group receiving Satisens® for 8 weeks, a placebo group, and a subgroup of the intervention group that will either continue with Satisens® or switch to placebo for an additional 4 weeks. The study uses a parallel assignment model to compare the effects of the intervention on emotional eating, appetite, and related biomarkers.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a double-blind study. Neither the participants nor the investigators will know whether the subject is receiving Satisens® or placebo. The placebo capsules are identical in appearance and administration schedule to the active product.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm 1: Satisens® 8 Weeks (Experimental): Participants receive 2 capsules of Satisens® daily for 8 weeks. The supplement contains lemon verbena, hibiscus, saffron, and other plant extracts. Capsules are taken with breakfast or lunch.
  Interventions: Dietary Supplement: Intervention 1: Satisens®
- Arm 1.1: Satisens® 12 Weeks (Experimental): Subgroup of Arm 1 continues with Satisens® for an additional 4 weeks (total 12 weeks). Same dosage and administration as initial 8 weeks.
  Interventions: Dietary Supplement: Intervention 1: Satisens®
- Arm 1.2: Satisens® 8 Weeks + Placebo 4 Weeks (Experimental): Subgroup of Arm 1 receives Satisens® for 8 weeks followed by placebo for 4 weeks. Placebo capsules are identical in appearance and administration.
  Interventions: Dietary Supplement: Intervention 1: Satisens®; Dietary Supplement: Intervention 2: Placebo
- Arm 2: Placebo 8 Weeks (Placebo Comparator): Participants receive placebo capsules for 8 weeks. Capsules are identical in appearance to Satisens® and contain inert ingredients.
  Interventions: Dietary Supplement: Intervention 2: Placebo

INTERVENTIONS:
Dietary Supplement: Intervention 1: Satisens® — A dietary supplement composed of lemon verbena (Lippia citriodora), hibiscus (Hibiscus sabdariffa), saffron (Crocus sativus), and carob extract. Administered as 2 capsules daily with breakfast or lunch. Used to modulate appetite, emotional eating, and inflammatory markers.
  Other Names: Satisens®; Plant-based satiety supplement
  Arms: Arm 1.1: Satisens® 12 Weeks; Arm 1.2: Satisens® 8 Weeks + Placebo 4 Weeks; Arm 1: Satisens® 8 Weeks
Dietary Supplement: Intervention 2: Placebo — Identical in appearance to the active supplement. Contains water with sucrose and no active ingredients. Administered as 2 capsules daily with breakfast or lunch.
  Other Names: Placebo capsule; Sucrose capsule
  Arms: Arm 1.2: Satisens® 8 Weeks + Placebo 4 Weeks; Arm 2: Placebo 8 Weeks

SUMMARY:
This study evaluates the efficacy of Satisens®, a dietary supplement composed of plant extracts, in reducing emotional eating and sweet cravings in healthy adults. The study will analyze hormonal, neurotransmitter, and inflammatory markers to understand the underlying mechanisms.

DETAILED DESCRIPTION:
This study aims to evaluate the efficacy of Satisens®, a dietary supplement composed of lemon verbena (Lippia citriodora), hibiscus (Hibiscus sabdariffa), and saffron (Crocus sativus), in reducing emotional eating and sweet cravings in healthy adults. The supplement is hypothesized to modulate appetite through neuroendocrine and anti-inflammatory mechanisms.

The study is a prospective, longitudinal, mixed-method, analytical, and experimental clinical trial. Participants will be randomly assigned to intervention or placebo groups. The intervention group will receive two capsules of Satisens® daily for 8 weeks, with a subgroup continuing for an additional 4 weeks or switching to placebo. The placebo group will receive identical capsules without active ingredients.

Primary outcomes include changes in emotional eating, appetite, sweet cravings, body weight, BMI, waist circumference, and waist-to-hip ratio. Secondary outcomes include blood levels of appetite-related hormones, neurotransmitters, and inflammatory markers.

Emotional eating will be assessed using validated questionnaires (EEQ, VAS, PFS). Blood samples will be analyzed using chromatography and mass spectrometry techniques. Statistical analysis will include paired t-tests or Wilcoxon tests, Mann-Whitney U tests, correlation analysis, and structural equation modeling.

The study has received ethical approval from the Ethics Committee of the Universidad Católica de Valencia San Vicente Mártir (code: UCV/2024-2025/015) and complies with the Declaration of Helsinki and GDPR regulations.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 65 years
* Healthy individuals without chronic diseases
* Able to provide informed consent

Exclusion Criteria:

* Pregnant or breastfeeding women
* Individuals taking medications or supplements that may interfere with study variables
* Individuals engaging in more than 3 hours of active exercise per week

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in Emotional Eating Score (EEQ) | Baseline, Week 8, Week 12
  Measured using the Emotional Eating Questionnaire (EEQ) to assess changes in emotional eating behavior.
  Scale Range: 0 to 30 Interpretation: Higher scores indicate worse emotional eating behavior (i.e., greater tendency to eat in response to emotions).
Change in Appetite Score (VAS) | Baseline, Week 8, Week 12
  Visual Analog Scale adapted for appetite, including hunger, satiety, fullness, and prospective food consumption.
  Scale Range: 0 to 100 for each item Interpretation: Higher scores indicate greater satiety and lower appetite. Therefore, a higher PA score reflects a better outcome in terms of appetite control.
Change in Sweet Craving (PFS) | Baseline, Week 8, Week 12
  Power of Food Scale adapted to sweet foods to assess psychological craving. Scale Range: 1 to 5 per item (typically 15 items total; total score range: 15 to 75) Interpretation: Higher scores indicate greater psychological craving for sweet foods, thus a worse outcome in the context of this study.
Change in Body Weight | Baseline, Week 8, Week 12
  Measured in kilograms (kg) using a calibrated scale with participants in a fasting state.
  Unit of Measure: Kilograms (kg) Interpretation: A decrease in weight indicates a better outcome.
Change in Body Mass Index (BMI) | Baseline, Week 8, Week 12
  Calculated as weight (kg) divided by height squared (m²). Unit of Measure: kg/m² Interpretation: A decrease in BMI indicates a better outcome.
Change in Waist Circumference | Baseline, Week 8, Week 12
  Measured in centimeters (cm) at the midpoint between the lower margin of the last palpable rib and the top of the iliac crest.
  Unit of Measure: Centimeters (cm) Interpretation: A decrease in waist circumference indicates a better outcome.
Change in Waist-to-Hip Ratio (WHR) | Baseline, Week 8, Week 12
  Calculated as waist circumference divided by hip circumference. Unit of Measure: Ratio (unitless) Interpretation: A decrease in WHR indicates a better outcome.

SECONDARY OUTCOMES:
Change in Appetite-Related Hormones | Baseline, Week 8, Week 12
  Blood levels of different Appetite-Related Hormones
Change in Neurotransmitter Levels | Baseline, Week 8, Week 12
  Blood levels of different Neurotransmitter
Change in Leptin Levels | Baseline, Week 8, Week 12
  Measured in serum using ELISA. Leptin is a hormone secreted by adipocytes that signals satiety to the hypothalamus.
  Unit of Measure: ng/mL Interpretation: A decrease in leptin levels (in the context of leptin resistance) may indicate improved sensitivity and better appetite regulation.
Change in Adiponectin Levels | Baseline, Week 8, Week 12
  Measured in serum using ELISA. Adiponectin is an anti-inflammatory adipokine associated with improved metabolic health and satiety.
  Unit of Measure: µg/mL Interpretation: An increase in adiponectin levels indicates a better outcome (improved metabolic and inflammatory profile).
Change in Ghrelin Levels | Baseline, Week 8, Week 12
  Measured in serum using ELISA. Ghrelin is known as the "hunger hormone" and stimulates appetite.
  Unit of Measure: pg/mL Interpretation: A decrease in ghrelin levels indicates a better outcome (reduced hunger signaling).
Change in Interleukin-6 (IL-6) Levels | Baseline, Week 8, Week 12
  Measured in serum using ELISA (Enzyme-Linked Immunosorbent Assay). Unit of Measure: pg/mL Interpretation: A decrease in IL-6 levels indicates a better outcome (reduced inflammation).
Change in Tumor Necrosis Factor-alpha (TNF-α) Levels | Baseline, Week 8, Week 12
  Measured in serum using ELISA (Enzyme-Linked Immunosorbent Assay). Unit of Measure: pg/mL Interpretation: A decrease in TNF-α levels indicates a better outcome (reduced inflammation).

CONTACTS AND LOCATIONS:
Overall Officials: José Enrique Dr. de la Rubia Ortí, PhD in Pharmacy, Principal Investigator — Universidad Católica de Valencia San Vicente Mártir; Gonzalo Mariscal Ruiz-Rico, Principal Investigator — Universidad Católica de Valencia San Vicente Mártir; Ana Belén Carriquí Suárez, Study Director — Facultad de Medicina y Ciencias de la Salud, Universidad Católica de Valencia
Locations (1):
- Universidad Católica de Valencia San Vicente Mártir - Facultad de Medicina y Ciencias de la Salud, Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to institutional data protection policies and the nature of the study, which involves sensitive health-related and psychological information. Data will be handled in compliance with the EU General Data Protection Regulation (GDPR) and Spanish data protection laws, and will remain confidential and accessible only to the research team.

REFERENCES:
- See also: Official website of Universidad Católica de Valencia San Vicente Mártir, where the study is being conducted. — https://www.ucv.es
- See also: Official profile of Dr. José Enrique de la Rubia Ortí and his research group "El estrés y la enfermedad" at the Catholic University of Valencia. Includes academic background, research lines, and scientific publications. — https://portalcientifico.ucv.es/es/ipublic/researcher/324253
- See also: Official website of IVB Wellness Lab, the company collaborating on the clinical trial. Founded by Dr. Isabel Viña Bas, the company develops scientifically backed nutritional supplements, including SatiSens. — https://ivbwellness.com
- See also: Official news release from the Catholic University of Valencia announcing the clinical trial on a saffron-based supplement aimed at reducing sweet cravings and emotional eating. — https://www.ucv.es/actualidad/todas-las-noticias/estudian-un-suplemento-a-base-de-azafran-para-combatir-los-antojos-dulces
- See also: Media article discussing the potential of the saffron-based supplement SatiSens as a natural alternative to appetite suppressants, highlighting its role in the clinical trial. — https://okdiario.com/salud/azafran-nuevo-ozempic-que-reduce-antojos-dulces-mejora-saciedad-14146516